CLINICAL TRIAL: NCT02047617
Title: Study of Safety and Efficacy on Neuromyopathy of Early Standing With the Assistance of Tilt Table in Critically Patients
Acronym: TILT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Chirurgical Marie Lannelongue (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: P12-37815003/2012A00665-38; IDRCB 2012-A00665-38 (Other: P12-37815003)
Record Dates: First submitted 2013-10-07; First posted 2014-01-28 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Patients Are Recruited From One Thoracic and Cardiac Surgery ICU
Keywords: Muscle Weakness; Exercise therapy; Physiotherapy; Critical illness; Intensive care; Mechanical ventilation; Rehabilitation
MeSH Terms: conditions — Muscle Weakness; Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- the standard physiotherapy group (Active Comparator): Physiotherapy rehabilitation techniques used in the management of this group include passive range of motion, active range of motion/bed exercises, sitting at edge of bed, sitting in armchair, active transfer from the bed to chair. Mobilization and rehabilitation program is progressively introduced after clinical stabilization with a goal of progressing to ambulation and pulmonary rehabilitation.
  Interventions: Device: the standard physiotherapy group
- standing table group (Experimental): The same program as standard physiotherapy group is applied, with daily sessions of standing table in supplement. Standing table was performed on a motorized tilt table (ref: table de verticalisation, Franco&fils). The protocol involved a stepwise process to gradually raise the subject into a standing position on the standing table platform, at 10° intervals from 30° to 80°.
  Interventions: Device: standing table group

INTERVENTIONS:
Device: the standard physiotherapy group — Mobilization and rehabilitation program is progressively introduced after clinical stabilization
  Arms: the standard physiotherapy group
Device: standing table group — The protocol involved a stepwise process to gradually raise the subject into a standing position on the standing table platform
  Arms: standing table group

SUMMARY:
Critically ill patients frequently develop muscle weakness due to critical illness-related acute neuropathy and/or myopathy. This disorder is associated with difficulties in weaning from mechanical ventilation, prolonged intensive care unit and hospital stay, and increased mortality rates. In addition, many patients continue to suffer from decreased exercise capacity and quality of life for months to years after the acute event.

Besides controlling risk factors, no specific prevention or treatment exists. Recommendations advice to start early with active and passive exercise in critically ill patients (1). Having critically ill patients alert and engaged in progressive rehabilitation leading to mobilization, despite the use of life support therapies may reduce muscle atrophy and lead to improved strength and physical function (2).

This randomized controlled trial was designed to investigate whether a daily training session using a tilt table, started early in stable critically ill patients with an expected prolonged ICU stay, could induce a beneficial effect on exercise performance, quadriceps force and functional autonomy at ICU and hospital discharge compared to a standard physiotherapy program.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had been intubated and mechanically ventilated for more than 3 days, without weaning of ventilation sheduled in 24 hours

Exclusion Criteria:

* Polytrauma,
* Cerebral , spinal cord or spinal injury,
* Pelvic or lower limb fracture

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2013-08; Primary Completion 2015-08 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Measure of overall muscle strength, a composite Medical Research Council score (MRC score) from examination of 3 muscle groups in each limb is used. | Medical Research Council, the patient is monitored and evaluate for up to 1 month
  Clinically important muscle weakness has been defined as a composite MRC score <80% of normal (eg, a score <48 out of a maximum of 60 based on examination of 3 muscle groups in each limb).
  MRC score is measured after randomization, before ICU discharge and before hospital discharge.

SECONDARY OUTCOMES:
The time to standing | Duration ( time and every day), the patient is monitored and evaluate for up to 1 month
  This secondary endpoint is measured every day until the leaving of ICU and continued until leaving the hospital.
ICU stay | duration (day number), the patient is monitored and evaluate for up to 1 month
Hospital stay | duration (day number), the patient is monitored and evaluate for up to 1 month
Mechanical ventilation duration | time in minutes (every day), the patient is monitored and evaluate for up to 1 month
  This secondary endpoint is measured every day until the leaving of ICU and continued until leaving the hospital.
Hospital mortality | number of death during the 3 years of the study
  number of deaths
Changes in blood pressure of more or less 20% of the reference value of rest required to stop the session or initiation of medical treatment | Blood Pressure(mm Hg) before and during standing session (every day). the patient is monitored and evaluate for up to 1 month
  This secondary endpoint is measured every day until the leaving of ICU and continued until leaving the hospital.
Changes in heart rate of more or less 20% of the reference value of rest required to stop the session or initiation of medical treatment | heartt rate (beats a minute) before and during standing session (every day). the patient is monitored and evaluate for up to 1 month
  This secondary endpoint is measured every day until the leaving of ICU and continued until leaving the hospital.
Onset of arrhythmia | irregular heart beat, every day the patient is monitored and evaluate for up to 1 month
  This secondary endpoint is measured every day until the leaving of ICU and continued until leaving the hospital.
Appearance of a disorder repolarization | ECG Interpretation, every day the patient is monitored and evaluate for up to 1 month
  This secondary endpoint is measured every day until the leaving of ICU and continued until leaving the hospital.
desaturation of more than 10% of the reference value requiring a decision of the meeting or any medical intervention, | % saturation, every day, the patient is monitored and evaluate for up to 1 month
  This secondary endpoint is measured every day until the leaving of ICU and continued until leaving the hospital.
Increase in systolic pulmonary artery pressure more than 60 mmHg | systolic pulmonary artery pressure (every day), the patient is monitored and evaluate for up to 1 month
  This secondary endpoint is measured every day until the leaving of ICU and continued until leaving the hospital.
Pneumothorax detected immediately after standing session | Chest radiography and clinical examination, every day the patient is monitored and evaluate for up to 1 month
  This secondary endpoint is measured every day until the leaving of ICU and continued until leaving the hospital.
Agitation requiring the increase of sedation or complicated tear gastric catheter probe or endotracheal tube, | observation evry day, the patient is monitored and evaluate for up to 1 month
  This secondary endpoint is measured every day until the leaving of ICU and continued until leaving the hospital.
Fall of the patient during a transfer | observation, every day the patient is monitored and evaluate for up to 1 month
  This secondary endpoint is measured every day until the leaving of ICU and continued until leaving the hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Céline SARFATI, physiotherapist, Principal Investigator — Centre Chirurgical Marie Lannelongue
Locations (1):
- Centre Chirurgical MarieLannelongue, Le Plessis-Robinson, Île-de-France Region, France

REFERENCES:
- [Background] Gosselink R, Bott J, Johnson M, Dean E, Nava S, Norrenberg M, Schonhofer B, Stiller K, van de Leur H, Vincent JL. Physiotherapy for adult patients with critical illness: recommendations of the European Respiratory Society and European Society of Intensive Care Medicine Task Force on Physiotherapy for Critically Ill Patients. Intensive Care Med. 2008 Jul;34(7):1188-99. doi: 10.1007/s00134-008-1026-7. Epub 2008 Feb 19. PMID 18283429
- [Background] Schweickert WD, Pohlman MC, Pohlman AS, Nigos C, Pawlik AJ, Esbrook CL, Spears L, Miller M, Franczyk M, Deprizio D, Schmidt GA, Bowman A, Barr R, McCallister KE, Hall JB, Kress JP. Early physical and occupational therapy in mechanically ventilated, critically ill patients: a randomised controlled trial. Lancet. 2009 May 30;373(9678):1874-82. doi: 10.1016/S0140-6736(09)60658-9. Epub 2009 May 14. PMID 19446324
- [Derived] Sarfati C, Moore A, Pilorge C, Amaru P, Mendialdua P, Rodet E, Stephan F, Rezaiguia-Delclaux S. Efficacy of early passive tilting in minimizing ICU-acquired weakness: A randomized controlled trial. J Crit Care. 2018 Aug;46:37-43. doi: 10.1016/j.jcrc.2018.03.031. Epub 2018 Apr 5. PMID 29660670